CLINICAL TRIAL: NCT01329679
Title: Effects of Single and Multiple Energy Shots on Blood Pressure and Electrocardiographic Parameters: A Randomized, Double Blind, Crossover, Placebo-controlled Trial
Brief Title: Impact of Energy Drinks on Cardiovascular Endpoints
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough subjects
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sachin Shah, Assistant Professor of Pharmacy Practice, David Grant U.S. Air Force Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FWH20110111H
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Energy Drinks; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy Drink (Experimental): Energy drink, 2 oz twice daily for 7 days
  Interventions: Dietary Supplement: Energy Drink
- Placebo (Placebo Comparator): Water, lime juice and cherry flavoring, 2 oz twice daily for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Energy Drink — Energy drink, 2oz twice daily for 7 days
  Arms: Energy Drink
Other: Placebo — Water, lime juice and cherry flavoring
  Other Names: Water, lime juice and cherry flavoring
  Arms: Placebo

SUMMARY:
Objective: To assess the cardiac effects of a an energy drink on blood pressure and heart rhythm in healthy subjects.

Study design: Double blind, placebo controlled, cross-over

Study population: Healthy human volunteers (active-duty) between age 18 to 40 years with no other medical conditions.

Intervention: Energy drink or Placebo

Primary outcome: Change in office systolic blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between ages 18-40 years
* ONLY "as needed" use of ibuprofen or acetamenophen
* Active duty military
* DoD beneficiary or Civilian Government Employees

Exclusion Criteria:

* No other co-morbid conditions
* No active prescription or OTC drug use
* Not pregnant or planning to become pregnant during study participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shah Sachin, Pharm.D., Principal Investigator — David Grant Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Energy Drink, Then Placebo: Energy drink, 2 oz twice daily for 7 days, washout period, then Placebo: Water, lime juice and cherry flavoring
- Placebo, Then Energy Drink: Placebo: Water, lime juice and cherry flavoring, 2 oz twice daily for 7 days, washout period, then energy drink, 2 oz twice daily for 7 days
Period: Overall Study
Arm/Group | Energy Drink, Then Placebo | Placebo, Then Energy Drink
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Energy drink: Energy drink, 2oz twice daily for 7 days Placebo: Water, lime juice and cherry flavoring
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 28.3 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20
  African American | 2
  Asian | 2
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Office Systolic Blood Pressure
Description: SBP = Systolic Blood Pressure measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days.
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
mmHg
  SBP at baseline | 128 (9.98) | 123 (8.49)
  SBP at Day 7 | 127 (9.88) | 124 (8.29)

2. Secondary Outcome: Office DBP After a Single Energy Shot and After Chronic Consumption
Description: DBP = Diastolic Blood Pressure measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days.
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
mmHg
  Baseline | 82.7 (7.79) | 79.0 (6.80)
  Day 7 | 82.2 (6.84) | 78.7 (6.33)

3. Secondary Outcome: Max Heart Rate After a Single Shot and After Chronic Consumption
Description: Maximum heart rate measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Energy Drink: Energy drink: Energy drink, 2 oz twice daily for 7 days
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
beats per minute
  Baseline | 69.8 (9.50) | 70.3 (8.41)
  Day 7 | 68.1 (9.21) | 67 (7.7)

4. Secondary Outcome: Max PR-interval After a Single Shot and After Chronic Consumption
Description: Maximum PR-interval measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
msec
  Baseline | 166 (18.8) | 161 (17.3)
  Day 7 | 164 (15) | 164 (16.7)

5. Secondary Outcome: Max QRS Duration After a Single Shot and After Chronic Consumption
Description: Max QRS duration measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
msec
  Baseline | 92.1 (9.18) | 92.3 (9.26)
  Day 7 | 94.8 (10.5) | 93.4 (8.76)

6. Secondary Outcome: Max QT Interval After a Single Energy Shot or Placebo Consumption After Day 1 and After Chronic Consumption After Day 7
Description: Max QT interval measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
msec
  Baseline | 414 (21.9) | 412 (16.2)
  Day 7 | 422 (21.2) | 418 (21)

7. Secondary Outcome: Max QTc Interval After a Single Energy Shot or Placebo Consumption After Day 1 and After Chronic Consumption After Day 7
Description: Max QTc interval measured at baseline (after a single energy shot or placebo consumption) and after chronic consumption for 7 days
Time Frame: At baseline and 7 days post energy drink and placebo consumption
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Energy Drink | Placebo
Number analyzed (Participants) | 26 | 26
msec
  Baseline | 422 (15.3) | 424 (18)
  Day 7 | 426 (20.1) | 419 (21.5)

ADVERSE EVENTS:
Time Frame: During the study, for up to 7 days per intervention
Arm/Group | Energy Drink | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
Small sample size and limited to 7 days of consumption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No